CLINICAL TRIAL: NCT04424784
Title: Influence of Manipulation of Oocytes and Embryos in Low Oxygen Tension on Assisted Reproduction Technology Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HKUSZH201902022
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Embryo Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% O2 (No Intervention): In the control group, oocyte pickup will be performed in atmospheric oxygen environment (20% oxygen, 89% nitrogen, 6% carbon dioxide).
- 5% O2 (Experimental): In the experimental group, oocyte pickup will be performed in a low oxygen tension environment (5% oxygen, 89% nitrogen, 6% carbon dioxide). If time lapse embryo culture system is used, fertilization check and embryo grading will also be conducted under the low oxygen tension environment.
  Interventions: Biological: 5% O2

INTERVENTIONS:
Biological: 5% O2 — 5% oxygen will be used during oocyte retrieval, fertilization check and embryo grading
  Arms: 5% O2

SUMMARY:
Nowadays, most assisted reproduction laboratories attempt to maintain as much as possible ex vivo culture conditions comparable to those in vivo. Various culturing condition such as temperature and pH parameters have been adjusted according to in vivo values in order to improve in-vitro fertilization (IVF) outcomes. Embryos of most mammals, including that of humans, are not exposed to oxygen concentration higher than 8%. Thus, embryos and gametes should be kept in a low oxygen environment during manipulation in assisted reproduction treatment.

Culturing embryos in low oxygen concentrations is now a general practice in IVF laboratories. However, there are still laboratory procedures when the oocytes/embryos are exposed to atmospheric oxygen. In most laboratories, oocytes retrieval is performed under atmospheric oxygen concentration. Oocyte is very sensitive to environmental changes, for instance, transient cooling to room temperature can cause irreversible disruption of the meiotic spindle in human oocytes and oocyte in vitro maturation can lead to the decline of energy metabolism in human oocytes. Whether oocyte exposed to atmospheric oxygen during oocyte retrieval has detrimental effect on embryo development and IVF outcomes is unknown.

Previous studies showed that low oxygen tension during embryo culture improved implantation rate and clinical outcomes, but embryo quality was not affected. In other studies, embryo quality was improved but overall pregnancy was not affected. The reason for the discrepancies could be because the oxygen tension during oocyte/embryo manipulation was not under well control. For instance, oocyte retrieval, fertilization check and embryo grading were performed under atmospheric oxygen. It is difficult to predict how these factors negatively impact the IVF outcomes.

In this project, the investigators hypothesize that lower oxygen tension during oocyte/embryo manipulation improves IVF outcomes.

DETAILED DESCRIPTION:
In the experimental group, oocyte pickup will be performed in a lower oxygen tension environment (5% oxygen, 89% nitrogen, 6% carbon dioxide); oocyte pickup will be performed in a special workstation with reduced oxygen tension environment while fertilization check and embryo grading will be performed in conventional and time lapse embryo culture system. The time lapse culture system can provide a constant lower oxygen tension culture environment to the embryos. In the control group, oocyte pickup, fertilization check and embryo grading will be performed in atmospheric oxygen environment. Under this arrangement, the difference between the 2 groups is the oxygen tension during oocyte/embryo manipulation. The investigators believe that a solid conclusion can be drawn about whether lower oxygen tension environment can benefit IVF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all the couples undergoing conventional IVF cycle in the reproductive medicine center of the University of Hong Kong-Shenzhen Hospital

Exclusion Criteria:

* Intracytoplasmic sperm injection (ICSI) cycle
* Preimplantation genetic testing (PGT) cycle
* cycle with fertilization failure ≥3
* cycle using sperm from percutaneous epididymal sperm aspiration (PESA)/testicular sperm extraction (TESE) or cryopreserved sperm
* cycle using cryopreserved oocyte
* cycle with no oocyte retrieved

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 4 years
  delivery of a live birth beyond 24 weeks of gestation

SECONDARY OUTCOMES:
clinical pregnancy rate | 3 years
  presence of at least one gestational sac on ultrasound of 6 weeks
ongoing pregnancy rate | 3 years
  presence of at least heart pulsation on ultrasound beyond 20 weeks
fertilization rate | 3 years
  No. of fertilized oocyte divided by No. of inseminated cumulus-oocyte complexes (COCs)
cleavage rate | 3 years
  No. of cleaved embryo divided by No. of fertilized oocyte

CONTACTS AND LOCATIONS:
Overall Officials: Shubiu Yeung, PhD, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (1):
- Reproductive medicine center, Shenzhen, China

REFERENCES:
- [Background] Fischer B, Bavister BD. Oxygen tension in the oviduct and uterus of rhesus monkeys, hamsters and rabbits. J Reprod Fertil. 1993 Nov;99(2):673-9. doi: 10.1530/jrf.0.0990673. PMID 8107053
- [Background] Kovacic B, Vlaisavljevic V. Influence of atmospheric versus reduced oxygen concentration on development of human blastocysts in vitro: a prospective study on sibling oocytes. Reprod Biomed Online. 2008 Aug;17(2):229-36. doi: 10.1016/s1472-6483(10)60199-x. PMID 18681997
- [Background] Waldenstrom U, Engstrom AB, Hellberg D, Nilsson S. Low-oxygen compared with high-oxygen atmosphere in blastocyst culture, a prospective randomized study. Fertil Steril. 2009 Jun;91(6):2461-5. doi: 10.1016/j.fertnstert.2008.03.051. Epub 2008 Jun 12. PMID 18554591